CLINICAL TRIAL: NCT03144128
Title: The Contribution of Vitamin D to Muscle Metabolic Function in Cancer Cachexia
Brief Title: Vitamin D for Muscle Metabolic Function in Cancer Cachexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Travis Thomas (Other)
Responsible Party: Sponsor-Investigator, David Travis Thomas, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MCC-15-LUN-102; MCC Protocol #15-1024-F1V (Other: Univ of KY Markey Cancer Center)
Record Dates: First submitted 2017-03-20; First posted 2017-05-08 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cancer Cachexia; Vitamin D Deficiency
Keywords: vitamin D; muscle; metabolism; cancer cachexia
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Prospective, double-blinded randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects receive exercise and protein supplementation. Participants, Investigators, Care Providers, and outcome assessors will be blinded to vitamin D vs. placebo capsule allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Ctl) (Placebo Comparator): Standard of Care resistance exercise and timed protein supplementation with placebo capsule daily for 12 weeks
  Interventions: Dietary Supplement: Placebo
- Vitamin D (Experimental): Standard of Care resistance exercise and timed protein supplementation with 5,000IU vitamin D supplementation daily for 12 weeks
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — 5,000IU vitamin D given daily for 12 weeks
  Arms: Vitamin D
Dietary Supplement: Placebo — Placebo capsules given daily for 12 weeks
  Arms: Control (Ctl)

SUMMARY:
The proposed study is aimed at examining mitochondrial function as a potential target of action of vitamin D on muscle metabolism, size, and strength in preventing the progression of cachexia. This is the first clinical trial designed to understand the effects of vitamin D on muscle metabolic dynamics driving dysfunction in cachectic muscle. Our preliminary data suggest that vitamin D promotes lipid partitioning and muscle metabolic function, which the investigators hypothesize, will mitigate cachexia via improved muscle health and quality that translates into reduced fatigue, and improved patient resilience to multimodal cancer therapy.

DETAILED DESCRIPTION:
Vitamin D repletion is linked to improved muscle mitochondrial function, lipid deposition and preservation; however, while vitamin D insufficiency is common in cancer, the mechanistic effects of vitamin D on muscle metabolic health in cancer patients have not been studied. This is important to address because cancer cachexia is characterized by marked muscle wasting, anabolic resistance, ectopic fat infiltration, mitochondrial dysfunction and contributes to decreased survival. With novel strategies to address this knowledge gap, the investigators will use a combination of advanced metabolic analytical approaches with complementary model systems in cell culture and human subjects to understand the biochemical and physiological mechanisms underlying cancer cachexia in relation to the role of vitamin D in conjunction with resistance exercise (RE). By combining analyses of muscle size and local tissue hemodynamics in vivo, metabolomics analyses of muscle tissue and isolated mitochondria, and changes in anabolic cell signaling, lipid metabolism and oxidative capacity of primary muscle cells in vitro, the investigators will identify mechanisms underlying muscle response to vitamin D repletion. Our previous findings, together with data that exercise improves muscle vitamin D storage and retrieval, suggest that vitamin D repletion synergizes with RE to improve muscle metabolic function and protein synthesis. Our overall objective is to examine mitochondrial function and anabolic resistance as potential targets of action of vitamin D on muscle metabolism, size and strength in preventing the progression of cachexia. The aims of this study are to: 1) non-invasively quantify lipid redistribution, local muscle tissue metabolism and muscle mass and strength of cancer patients before and after 12 weeks of double blinded vitamin D repletion with exercise and protein supplementation (VitD) compared to exercise and protein supplementation only (Ctl); 2) determine differences in muscle mitochondrial function in live tissue biopsied from human gastrocnemius from VitD compared to Ctl; and 3) identify mechanisms whereby vitamin D and exercise regulate muscle anabolic signaling and mitochondrial activity in primary human myotube cultures. Our central hypothesis is that vitamin D promotes muscle lipid availability for β-oxidation in response to exercise, thereby preventing lipotoxicity in the muscle and potentially improving anabolic sensitivity in muscle during cancer cachexia. The impact of this project, the first nutrition and exercise study designed as an inexpensive intervention, is to understand the effect of vitamin D on the metabolic and anabolic dynamics which underpin dysfunction in cachectic muscle. If vitamin D promotes lipid partitioning, muscle metabolic function and/or anabolic sensitivity, these adaptations will ultimately improve cancer therapy by combating cancer cachexia. Further, diffuse optical spectroscopy techniques have the potential to identify the minimum effective intervention dose for optimizing metabolic health leading to more practical and individualized lifestyle prescriptions to reduce health care costs.

ELIGIBILITY:
Inclusion Criteria:

Patients must have histologically or cytologically confirmed stage II-IV lung cancer and be planned for definitive non-surgical therapy.

Patients may have a history of prior malignancy.

Mild cancer cachexia, defined by the miniCASCO score of 0-25 points

Vitamin D insufficiency, defined as 25(OH)D < 32 ng/ml

Aged 45 to 75 years. Stratified randomization by age

ECOG performance status ≤ 2 (see Appendix A).

Life expectancy of greater than 3 months

Patients must have normal renal and liver function as defined below:

AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal creatinine within normal institutional limits OR creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

Able to swallow thin liquids

No uncontrolled illness including, but not limited to, any of the following:

* Ongoing or active serious infection
* Symptomatic congestive heart failure
* Unstable angina pectoris
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension
* Psychiatric illness or social situation that would preclude compliance with study requirements

Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.

Patients with untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with treated brain metastasis are eligible for this trial, providing they have completed treatment at least one day prior to registration.

History of allergic reactions to whey or milk proteins.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Patients with a history of calcium oxalate nephrolithiasis are excluded.

Patients with a significant history of malabsorption (e.g. celiac sprue, short bowel syndrome, IBD or other, as determined by the treating physician) are excluded.

Patients will not be eligible if actively receiving treatment for vitamin D deficiency and have had recent (3 month) history of vitamin D supplementation (>1000 IU) or calcium supplementation (>800mg).

The following exclusion criteria will avoid the possibility of preexisting muscle impairment: history of congenital myopathies; neurologic disorder involving sequelae of spinal derangement; disk disease or vascular disease; tremor and rigidity.

Patients will also be excluded if they report lower extremity (LE) surgery or injury to the LE in the past 3 months or a past medical history of primary hyperparathyroidism; or rhabdomyolysis.

Additional exclusion criteria include participation in a scheduled resistance exercise program 1 month;

* metal implants or other contraindications for the MRI;
* diabetes,
* advanced renal disease,
* uncontrolled hypertension;
* a vitamin D status (25(OH)D) of > 32ng/mL.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Non-invasive quantification of muscle lipid distribution | Change between Week 0 and Week 12
  MRI/MRS
Local muscle oxygen consumption | Change between Week 0 and Week 12
  Near Infrared Spectroscopy + Diffuse Correlation Spectroscopy measures will be combined to assess changes in local muscle tissue oxygen consumption (VO2 measure)
Muscle Mass | Change between Week 0 and Week 12
  MRI
Muscle Strength | Change between Week 0, Week 6, Week 12
  Maximal voluntary contractions and 1-Repetition Maximum will be aggregated to to provide a comprehensive assessment of muscle strength

SECONDARY OUTCOMES:
Mitochondrial Function in Muscle Fibers in Fresh Muscle Fibers ex vivo | Experiments will be conducted from tissue collected at week 12 study biopsy
  Determine the differences in muscle mitochondrial function in live tissue biopsied from human gastrocnemius from VitD compared to Ctl by measure live tissue oxygen consumption rate. Respiration measures will be combined to assess mitochondrial function
  Mitochondrial respiration will be measured by the XF96 Seahorse extracellular flux analyzer
Mitochondrial Function in Muscle Fibers in Fresh Muscle Fibers ex vivo | Experiments will be conducted from tissue collected at week 12 study biopsy
  Determine the differences in muscle mitochondrial function in live tissue biopsied from human gastrocnemius from VitD compared to Ctl by measure live tissue oxygen consumption rate. Fatty acid oxidation measures will be combined to assess mitochondrial function
  Fatty acid oxidation will be estimated by monitoring the OCR of cells with no exogenous glucose or glutamine (Gln) ± a specific fatty acid oxidation (FAO) inhibitor, etomoxir (40 µM)
Stable Isotope-Resolved Metabolomics to describe Fatty Acid Metabolism in relationship to other fuel substrates in Fresh Muscle Fibers ex vivo | Experiments will be conducted from live tissue collected at week 12 study biopsy
  Determine the relative importance of vitamin D on lipid, amino acid and energy metabolism involving glucose, glutamine, and β-oxidation in intact muscle fibers. We will culture with 13C8-octanoate, 13C6-glucose, or 13C5-Gln and measure metabolite isotopomer distributions to accomplish this goal.
Utilize cell culture experimentation to understand anabolic signaling in response to vitamin D with or without fiber stretch. | Experiments will be conducted from tissue collected at week 12 study biopsy
  Identify mechanisms whereby vitamin D and RE regulate anabolic signaling in primary human myotube cultures. Changes in signaling pathways associated with hypertrophy, including Akt, mTOR, MAPK, and AMPK, will be measured by phospho-western blot to determine response to calcitriol, palmitate, and stretch treatment in myotubes.
Utilize cell culture experimentation to measure mitochondrial activity in response to vitamin D with or without fiber stretch. | Experiments will be conducted from tissue collected at week 12 study biopsy
  To understand how vitamin D and RE regulate mitochondrial activity in primary human myotube cultures, the investigators will measure extracellular acidification rate (ECAR) in response to calcitriol supplementation. This will be assessed through the addition of CPT-1 inhibitor etomoxir (40 µM) and the ATP-synthase inhibitor oligomycin
Utilize cell culture experimentation to measure mitochondrial activity in response to vitamin D with or without fiber stretch. | Experiments will be conducted from tissue collected at week 12 study biopsy
  Identify mechanisms whereby vitamin D and RE regulate mitochondrial activity in primary human myotube cultures.
  The investigators will measure the concentration of ATP in myotubes in response to calcitriol supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No